CLINICAL TRIAL: NCT02675881
Title: Monopolar Radiofrequency Ablation Using a Dual Switching System and a Separable Clustered Electrode (Octopus®) for Treatment of Focal Liver Malignancies: A Preliminary Study
Brief Title: Monopolar Radiofrequency Ablation Using a Dual Switching System and a Separable Clustered Electrode (Octopus®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-2013-1441
Record Dates: First submitted 2016-01-31; First posted 2016-02-05 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: HCC; Metastasis
Keywords: RFA
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA DSM (Active Comparator): Eligible patients who undergo RFA using DSM and separable clustered electrodes.
  Interventions: Device: DSM; Device: separable clustered electrode
- RFA SSM (No Intervention): Historical control group consisted of patients underwent RFA in our institution with single switching mode (SSM) and single/ or multiple clustered electrodes.

INTERVENTIONS:
Device: DSM — Monopolar RFA using dual switching mode (DSM)
  Arms: RFA DSM
Device: separable clustered electrode — A separable clustered electrode is similar to a clustered electrode, although it differs from a conventional clustered electrode in that each individual electrode is separable.
  Other Names: Octopus(R)
  Arms: RFA DSM

SUMMARY:
Increasing ablative zone is an essential part to improve technical success and long term outcome in patient treated with radiofrequency ablation (RFA).

A combination of dual switching system and separable clustered electrode has been reported to create large ablative zone in preclinical study.

Based on preclinical study, the investigators conducted a preliminary study in eligible 60 patients to measure whether this combination (dual switching system and separable clustered electrode) improves technical success rate and local tumor progression rate over a year, in comparison with historical control group.

DETAILED DESCRIPTION:
Increasing ablative zone is an essential part to improve technical success and long term outcome in patient treated with radiofrequency ablation (RFA).

A combination of dual switching system and separable clustered electrode has been reported to create large ablative zone in preclinical study.

Based on preclinical study, the investigators conducted a preliminary study in eligible 60 patients to measure whether this combination (dual switching system and separable clustered electrode) improves technical success rate and local tumor progression rate over a year, in comparison with historical control group using propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (according to AASLD guideline or LI-RADS)
* histologically confirmed HCC
* histologically confirmed or typical imaging feature of colorectal cancer liver metastasis in patients with colorectal cancer AND
* equal to or larger than 2cm, equal to or smaller than 5cm
* available cross-sectional liver imaging within 30 days before RFA
* signed informed consent

Exclusion Criteria:

* history of local treatment on the index tumor
* more than three tumors in a patient
* tumors in central portion of portal vein or hepatic vein
* Child-Pugh class C
* vascular invasion by tumors
* uncorrected coagulopathy
* presence of multiple extrahepatic metastases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2015-04-08 (Actual); Study Completion 2015-07-13 (Actual)

PRIMARY OUTCOMES:
local tumor progression (LTP) | 12 months

SECONDARY OUTCOMES:
Technical success on 1 months follow-up imaging after RFA (no residual/progressed tumor) | 1 months
rate of intrahepatic distant recurrence (IDR) after RFA | 12 months
rate of extrahepatic metastasis (EM) after RFA | 12 months

OTHER OUTCOMES:
Number of complication of RFA | 6 months
  incidence of any possible complication related with RFA
Maximal diameter of ablative zone | 7 day
  Maximal diameter of ablative zone on post-RFA CT or MRI in a mm.
ablation time | 1 day
  ablation time in a patient
Real time US fusion image feasibility | 1 day after RFA procedure
  success or failure of accurate fusion between US and pre-RFA cross sectional images
Immediate evaluation of ablative zone via visual assess and pre-and post-RFA images registration. | 12 months
  Prediction of LTP by classifying patients according to assessing ablative margin in each method on a four point scale (1: residual tumor, 4: ablative margin equal to or larger than 5mm)
Volume of ablative zone | 7 days
  Volume of ablative zone on post-RFA CT or MRI in a mm3.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes